CLINICAL TRIAL: NCT03106220
Title: Exercise Intervention and Its Impact on Hospitalization - a Mulitcentered Study
Brief Title: Exercise Intervention - and Impact on Hospitalization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow patient accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kymberly D. Watt, MD, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 16-010102
Record Dates: First submitted 2017-03-30; First posted 2017-04-10 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Sarcopenia; Debility Due to Disease
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: home exercise vs standard care with cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home exercise (Active Comparator): participate in home exercise program
  Interventions: Behavioral: exercise
- standard care (Placebo Comparator): encouraged to join physical therapy and walking goals
  Interventions: Other: placebo

INTERVENTIONS:
Behavioral: exercise — home exercise program
  Arms: home exercise
Other: placebo — encourage walking and physical therapy per standard care.
  Arms: standard care

SUMMARY:
Skeletal muscle abnormalities (sarcopenia) and frailty are common complications seen in patients with end-stage liver disease. The presence of these complications portends poor prognosis. The purpose of this study is to assess the impact of a formal home based video strengthening program (REST) on sarcopenia and frailty. We also want to assess the impact of this exercise program on complication rates, hospitalization, on quality of life (QOL) and on survival.

ELIGIBILITY:
inclusion= waitlisted for liver transplant with poor 6MWT

Exclusion criteria include: age < 18 years, recent hospitalization (within 14 days) due to decompensation, variceal bleeding in the previous 1 month, large esophageal varices without primary prophylaxis, active excessive alcohol intake (in the previous 3 months), current overt uncontrolled hepatic encephalopathy, hepatopulmonary syndrome with uncontrolled hypoxia, portopulmonary hypertension, inability to perform exercise, or marked symptomatic comorbidities (cardiac, pulmonary, renal). multiorgan transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
6MWT | 3 months
  6 minute walk
hand grip | 3 months
  hand grip

CONTACTS AND LOCATIONS:
Overall Officials: Kymberly D Watt, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials